CLINICAL TRIAL: NCT02490046
Title: Single Centre Open-label Feasibility Study Evaluating the Use of D-mannose in Multiple Sclerosis
Brief Title: D-mannose for the Prevention of UTIs in Multiple Sclerosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: UCLH (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 14/0384
Record Dates: First submitted 2015-04-28; First posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Multiple Sclerosis; Recurrent Urinary Tract Infections
Keywords: D mannose; multiple sclerosis; recurrent urinary infections
MeSH Terms: conditions — Multiple Sclerosis; Urinary Tract Infections | interventions — Mannose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MS and rec UTIs not using a catheter (Experimental): people with multiple sclerosis and recurrent urinary tract infections with spontaneous voiding Intervention- will be given D-mannose
  Interventions: Dietary Supplement: D Mannose
- MS and rec UTIs using a catheter (Experimental): people with multiple sclerosis and recurrent urinary tract infections using either urethral or suprapubic indwelling catheter or intermittent catheterisation Intervention- will be given D-mannose
  Interventions: Dietary Supplement: D Mannose

INTERVENTIONS:
Dietary Supplement: D Mannose — Patients in both arms will receive D-mannose powder to be used 1.5 gm (one level-teaspoon) twice daily, to be added to any beverage, for 16 weeks.

SUMMARY:
This is a study to explore the feasibility of using D-mannose, a commonly used food supplement, in persons with multiple sclerosis reporting recurrent urinary tract infections. Twenty persons with multiple sclerosis (10 patients using catheters and 10 not using catheters) reporting recurrent urinary tract infections will receive D-mannose 1.5 grams twice daily for 16 weeks duration.

This will be explored through:

1. Assessing compliance to a 16-week course of D-mannose
2. Quantifying the number of prescriptions for antibiotics during the 16 weeks course of D-mannose

DETAILED DESCRIPTION:
Informed consent procedure: Potential participants will be approached in clinic and given a patient information sheet and adequate time will be given for the individual to read through the patient information sheet and for clarification of any queries or concerns. Informed consent will be obtained by one of the investigators involved in the conduct of the study prior to participation in the trial, following adequate explanation of the aims, methods, anticipated benefits and potential hazards of the study.

Screening Period: Before any screening procedures occur, participants will sign an Informed Consent Form.

During the screening evaluation the following procedures will be conducted and recorded for all patients:

* Informed Consent
* Evaluation of compliance with inclusion and exclusion criteria
* Demography and Past Medical History
* Vital signs including weight
* Physical examination including neurological examination
* Review of concomitant medications

Baseline assessments: A urine sample will be tested for an infection using Urine multistix in the Department of Uro-neurology, which is a routine clinical practice. Participants will enter a discussion about the symptoms of a urinary tract infection and be taught the use of Urine multistix. They will complete standardised validated questionnaires for overactive bladder syndrome (ICIQ-OAB, sf-Qualiveen® and EQ5D-5L™).

Treatment procedures: Patients will receive D-mannose powder to be used 1.5 gm (one level-teaspoon) twice daily, to be added to any beverage, for 16 weeks. D-mannose is classed as a food supplement and is widely available in the United Kingdom for purchase. D-Mannose will be sourced from D-Mannose Limited.

Subsequent assessments: Compliance will be assessed by using a Usage diary, on which the use of D-mannose will be marked and any problems noted. Acceptability and tolerability to D-mannose will be assessed through the diary. Additionally, patients will be phoned after one week, and after 8 weeks, to enquire about well-being and compliance.

Participants will be asked to note the number of prescriptions they receive during the 16 week course in a urinary tract infection diary. Suspected self-reported urinary tract infections will be noted in a diary, as well as the results of the urine multistix. Standard clinical practice will be followed and participants with a suspected urinary tract infection will inform their general practitionner, mid-stream urine samples sent to the lab and antibiotic treatment started. Patients will continue to take D-mannose. The usage diary has to be sent by the patients every week.

At week 16, patients will be asked to return for a second visit. Compliance and urinary tract infection diaries will be collected and reviewed. They will be asked to complete questionnaires (ICIQ-OAB, sf-Qualiveen® and EQ5D-5L™) and neurological status will be evaluated.

The study will be conducted in accordance with the International Conference on Harmonization Good Clinical Practice guidelines and the Declaration of Helsinki, and within local laws and regulations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a known diagnosis of Multiple sclerosis (all stages) who have been clinically stable for at least three months and reporting lower urinary tract symptoms.
2. Patient with recurrent urinary tract infections, defined as having at least two urinary tract infections in the preceding six months or three or more urinary tract infections in the preceding one year. Urinary tract infections were defined retrospectively by patient self-report and confirmation by urine culture.
3. Age over 18 years and below 65
4. Females of childbearing potential using effective contraception if sexually active - oral contraceptive pill (> 3 months use), condoms, intrauterine contraceptive device, depot injection

Exclusion Criteria:

1. Pregnancy or planning pregnancy
2. Breastfeeding
3. History of congenital urinary tract anomalies or interstitial cystitis
4. History of diabetes mellitus
5. Receiving antibiotic prophylaxis or cranberry extract preparations
6. Current urinary tract infection
7. Current vaginal infection
8. Any known allergies to D-mannose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-10 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Compliance (self-usage diary and weight of returned containers of D-mannose) | 16 weeks
  Compliance to a 16-week course of D-mannose as assessed using a self-usage diary and weight of returned containers of D-mannose. The number of days the participant does not use D-mannose and reasons for non-use will be noted.

SECONDARY OUTCOMES:
Antibiotic prescription (Number of prescriptions for antibiotics required) | 16 weeks
  Number of prescriptions for antibiotics required during the 16-week course

CONTACTS AND LOCATIONS:
Overall Officials: Jalesh Panicker, MD,FRCP, Principal Investigator — UCLH NHS Foundation Trust
Locations (1):
- The National Hospital for Neurology and Neurosurgery, London, United Kingdom

REFERENCES:
- [Background] Nakipoglu GF, Kaya AZ, Orhan G, Tezen O, Tunc H, Ozgirgin N, Ak F. Urinary dysfunction in multiple sclerosis. J Clin Neurosci. 2009 Oct;16(10):1321-4. doi: 10.1016/j.jocn.2008.12.012. Epub 2009 Jun 27. PMID 19560927
- [Background] de Seze M, Ruffion A, Denys P, Joseph PA, Perrouin-Verbe B; GENULF. The neurogenic bladder in multiple sclerosis: review of the literature and proposal of management guidelines. Mult Scler. 2007 Aug;13(7):915-28. doi: 10.1177/1352458506075651. Epub 2007 Mar 15. PMID 17881401
- [Background] The prevention and management of urinary tract infections among people with spinal cord injuries. National Institute on Disability and Rehabilitation Research Consensus Statement. January 27-29, 1992. J Am Paraplegia Soc. 1992 Jul;15(3):194-204. doi: 10.1080/01952307.1992.11735873. PMID 1500945
- [Background] Hoffman JM, Wadhwani R, Kelly E, Dixit B, Cardenas DD. Nitrite and leukocyte dipstick testing for urinary tract infection in individuals with spinal cord injury. J Spinal Cord Med. 2004;27(2):128-32. doi: 10.1080/10790268.2004.11753743. PMID 15162883
- [Background] Stohrer M, Blok B, Castro-Diaz D, Chartier-Kastler E, Del Popolo G, Kramer G, Pannek J, Radziszewski P, Wyndaele JJ. EAU guidelines on neurogenic lower urinary tract dysfunction. Eur Urol. 2009 Jul;56(1):81-8. doi: 10.1016/j.eururo.2009.04.028. Epub 2009 Apr 21. PMID 19403235
- [Background] Fowler CJ, Panicker JN, Drake M, Harris C, Harrison SC, Kirby M, Lucas M, Macleod N, Mangnall J, North A, Porter B, Reid S, Russell N, Watkiss K, Wells M. A UK consensus on the management of the bladder in multiple sclerosis. J Neurol Neurosurg Psychiatry. 2009 May;80(5):470-7. doi: 10.1136/jnnp.2008.159178. PMID 19372287
- [Background] Leary SM, Porter B, Thompson AJ. Multiple sclerosis: diagnosis and the management of acute relapses. Postgrad Med J. 2005 May;81(955):302-8. doi: 10.1136/pgmj.2004.029413. PMID 15879043
- [Background] Hennessey A, Robertson NP, Swingler R, Compston DA. Urinary, faecal and sexual dysfunction in patients with multiple sclerosis. J Neurol. 1999 Nov;246(11):1027-32. doi: 10.1007/s004150050508. PMID 10631634
- [Background] Correale J, Fiol M, Gilmore W. The risk of relapses in multiple sclerosis during systemic infections. Neurology. 2006 Aug 22;67(4):652-9. doi: 10.1212/01.wnl.0000233834.09743.3b. Epub 2006 Jul 26. PMID 16870812
- [Background] Buljevac D, Flach HZ, Hop WC, Hijdra D, Laman JD, Savelkoul HF, van Der Meche FG, van Doorn PA, Hintzen RQ. Prospective study on the relationship between infections and multiple sclerosis exacerbations. Brain. 2002 May;125(Pt 5):952-60. doi: 10.1093/brain/awf098. PMID 11960885
- [Background] Rakusa M, Murphy O, McIntyre L, Porter B, Panicker J, Fowler C, Scott G, Chataway J. Testing for urinary tract colonization before high-dose corticosteroid treatment in acute multiple sclerosis relapses: prospective algorithm validation. Eur J Neurol. 2013 Mar;20(3):448-452. doi: 10.1111/j.1468-1331.2012.03806.x. Epub 2012 Jul 21. PMID 22816507
- [Background] Everaert K, Lumen N, Kerckhaert W, Willaert P, van Driel M. Urinary tract infections in spinal cord injury: prevention and treatment guidelines. Acta Clin Belg. 2009 Jul-Aug;64(4):335-40. doi: 10.1179/acb.2009.052. PMID 19810421
- [Background] Jepson RG, Williams G, Craig JC. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD001321. doi: 10.1002/14651858.CD001321.pub5. PMID 23076891
- [Background] Gallien P, Amarenco G, Benoit N, Bonniaud V, Donze C, Kerdraon J, de Seze M, Denys P, Renault A, Naudet F, Reymann JM. Cranberry versus placebo in the prevention of urinary infections in multiple sclerosis: a multicenter, randomized, placebo-controlled, double-blind trial. Mult Scler. 2014 Aug;20(9):1252-9. doi: 10.1177/1352458513517592. Epub 2014 Jan 8. PMID 24402038
- [Background] Michaels EK, Chmiel JS, Plotkin BJ, Schaeffer AJ. Effect of D-mannose and D-glucose on Escherichia coli bacteriuria in rats. Urol Res. 1983;11(2):97-102. doi: 10.1007/BF00256954. PMID 6346629
- [Background] Kranjcec B, Papes D, Altarac S. D-mannose powder for prophylaxis of recurrent urinary tract infections in women: a randomized clinical trial. World J Urol. 2014 Feb;32(1):79-84. doi: 10.1007/s00345-013-1091-6. Epub 2013 Apr 30. PMID 23633128
- [Result] Compston A, Coles A. Multiple sclerosis. Lancet. 2002 Apr 6;359(9313):1221-31. doi: 10.1016/S0140-6736(02)08220-X. PMID 11955556
- [Result] Marrie RA, Cutter G, Tyry T, Vollmer T, Campagnolo D. Disparities in the management of multiple sclerosis-related bladder symptoms. Neurology. 2007 Jun 5;68(23):1971-8. doi: 10.1212/01.wnl.0000264416.53077.8b. PMID 17548546
- [Derived] Phe V, Pakzad M, Haslam C, Gonzales G, Curtis C, Porter B, Chataway J, Panicker JN. Open label feasibility study evaluating D-mannose combined with home-based monitoring of suspected urinary tract infections in patients with multiple sclerosis. Neurourol Urodyn. 2017 Sep;36(7):1770-1775. doi: 10.1002/nau.23173. Epub 2016 Nov 4. PMID 27813195